CLINICAL TRIAL: NCT04747145
Title: A Phase II Study Analyzing Pulsed Reduced Dose Radiotherapy in Upfront Glioblastoma (PRORADGLIO Study)
Brief Title: Analyzing Pulsed Reduced Dose Radiotherapy in Upfront Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael Straza, MD, PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00039277
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
Keywords: pulsed reduced dose radiotherapy; glioblastoma; pRDR
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pulsed reduced dose-rate radiotherapy (Experimental): Chemoradiation, adjuvant chemotherapy.
  Interventions: Device: Radiation; Drug: Concurrent Chemotherapy (Temozolomide); Drug: Adjuvant Chemotherapy (Temozolomide)

INTERVENTIONS:
Device: Radiation — 60 Gy to be delivered over 30 daily treatments in six weeks. Chemoradiation is to start no sooner than 3 weeks after surgery and not later than 8 weeks.
  Other Names: Pulsed Reduced Dose Radiotherapy; pRDR
Drug: Concurrent Chemotherapy (Temozolomide) — 75mg/m^2 x 42 days (concurrent chemotherapy with radiation). Chemoradiation is to start no sooner than 3 weeks after surgery and not later than 8 weeks.
  Other Names: TMZ; Temodar
Drug: Adjuvant Chemotherapy (Temozolomide) — Starting no sooner than 4 weeks after completion of chemoradiation, 150-200mg/m^2, days 1-5 of 28-day cycle, for minimum of six cycles and up to 12 cycles.
  Other Names: TMZ; Temodar

SUMMARY:
The primary protocol objective is to assess the impact of substituting pulsed reduced dose radiotherapy (pRDR) for standard radiation therapy in the upfront treatment of glioblastoma (GBM) on disease progression.

DETAILED DESCRIPTION:
This is a single-arm, single-center phase 2 study designed to assess the efficacy of pulsed reduced dose-rate radiotherapy in the initial treatment of maximally safely resected glioblastoma. The primary endpoint will be progression-free survival at six months. Patients with pathologically confirmed GBM who are planned for six weeks of adjuvant chemoradiation followed by six to12 months of adjuvant chemotherapy will be screened and enrolled after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study-related procedure that is not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Female or male subjects ≥ 18 years old at the time of informed consent.
3. Histologically confirmed new diagnosis of GBM according to updated World Health Organization (WHO) classification criteria.
4. Supratentorial tumor location.
5. Recovered from maximal debulking surgery, if applicable (gross total resection, partial resection and biopsy-only patients are all acceptable).
6. Planned for standard adjuvant chemoradiotherapy of approximately 60 Gy of radiation therapy (RT) , or biologically equivalent dose, according to local practice, and concomitant TMZ chemotherapy (75 mg/m^2 daily) Any other cytotoxic or biologic antitumor therapy received prior to enrollment will be considered an exclusion.
7. Planned treatment with adjuvant/maintenance TMZ (150 to 200 mg/m^2 daily x 5 d, q 28 days).
8. All patients with sufficient tissue must have had tissue submitted for O6-Methylguanine-DNA Methyltransferase (MGMT) promoter methylation determination prior to enrollment.
9. Karnofsky Performance Status Scale ≥ 70.
10. Life expectancy greater than at least three months.
11. Study start date at least three weeks out from brain surgery.
12. Stable or decreasing dose of corticosteroids for the last seven days prior to enrollment, if applicable.
13. Complete blood count (CBC) /differential obtained within 28 days prior to registration, with adequate bone marrow function defined as follows: absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3; platelets ≥ 100,000 cells/mm^3; hemoglobin ≥ 10.0 g/dL. (Note: the use of transfusion or other intervention to achieve Hgb ≥10.0 g/dL is acceptable.)
14. Female subjects who:

    1. Are postmenopausal for at least one year before the screening visit, OR
    2. Are surgically sterile, OR

    If they are of childbearing potential:

    i. Agree to practice one highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through four months after the last study intervention (female and male condoms should not be used together), OR ii. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
15. Male subjects, even if surgically sterilized (i.e., status postvasectomy), who:

    1. Agree to practice effective barrier contraception during the entire study treatment period from the time of signing the informed consent through four months after the last study intervention (female and male condoms should not be used together), OR
    2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

Exclusion Criteria:

1. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of three years. (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
2. Recurrent or multifocal malignant gliomas.
3. Any site of distant disease (i.e., leptomeningeal disease or drop metastases from the GBM tumor site).
4. Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields.
5. Severe, active comorbidity, defined as follows:

   * Unstable angina at registration.
   * Transmural myocardial infarction within the last six months prior to registration.
   * Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of ≥ 2 mm using the analysis of an EKG performed within 28 days prior to registration. (Note: EKG to be performed only if clinical suspicion of cardiac issue.)
   * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to.
   * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.
   * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration.
   * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.
   * End-stage renal disease (i.e., on dialysis or dialysis has been recommended).
6. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
7. Patents treated on any other therapeutic clinical protocols within 30 days prior to registration.
8. Inability to undergo MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Six months
  This outcome measure is the number of subjects whose disease has not progressed using the Macdonald Response Criteria, which has the following classifications: complete response, partial response, stable disease and progression.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Straza, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No